CLINICAL TRIAL: NCT05547113
Title: Vestibular Function and Quality of Life in Patients After Cochlear Implantation
Brief Title: Vestibular Function in Cochlear Implant Patients
Status: Recruiting | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Collaborators: University Hospital, Motol (Other)
Responsible Party: Principal Investigator, Sara Koutna, Principal Investigator, Charles University, Czech Republic
Other Study IDs: 323721
Record Dates: First submitted 2022-08-31; First posted 2022-09-21 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Cochlear Implantation
Keywords: vestibular function; cochlear implantation; postural stability

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cochlear implant patients: The group of patients will consist of 40 adult patients indicated for cochlear implantation at the Department of ENT and Head and Neck Surgery, 1st Faculty of Medicine and FN Motol. Patients who meet the indication criteria for implantation also meet the conditions for inclusion in the study, another criterias are absence of diseases of the bearing joints, absence of diseases peripheral nervous system or muscle disease and absence of disease vision that would prevent visual fixation.
  Interventions: Diagnostic Test: posturography

INTERVENTIONS:
Diagnostic Test: posturography — In our stabilometric laboratory we use for the posturography two Kistler stabilometric platforms (type 5619A, Switzerland) along with MARS software (version 5.0, Switzerland). We use the SYNAPSIS Subjective Vertical device (version 1.3.2, France) to examine the perception of the subjective visual vertical. The patients should also full fill 5 questionnaires to subjective evaluation of non-vestibular symptoms within ADL and QoL, namely for difficulties related to dizziness, tinnitus, orofacial function disorders and the occurrence of anxiety and depression. For this purpose we use Dizziness Handicap Inventory, Tinnitus Handicap Inventory, Facial Disability Index, Beck's Anxiety Inventory and Beck's Depression Inventory.
  Other Names: subjective visual vertical; questionnaires

SUMMARY:
A hearing loss is condition which significantly affects the quality of life. The prevalence of the hearing disorders is relatively high due to many conditions which may result in a deafness. In those cases where hearing aids are not a sufficient solution to these difficulties, cochlear implantation is the standard treatment. It has been more than 30 years since the first implantation in the Czech Republic. These days it is common surgical procedure for adults and even children and it replaces, at least in part, the function of the hair cells that are no longer able to stimulate the primary auditory neurons.. Recent studies have reported that cochlear implant does not affect only hearing, but also other functions of the inner ear - the vestibular system resulting in stability and spatial orientation. Postural control is provided by coordination of movement strategies and sensory functions. If one ore more of these components are compromised postural instability appears. Instability is one of the most common causes of reduced quality of life. The deaf are characterized by their compensatory mechanisms, where visual system dominates over somatosensory and vestibular. After the cochlear implantation the postural behavior and compensations are changing apparently. The investigators assume that these mechanisms can be affected by vestibular rehabilitation. The purpose of this projet, will be to evaluate whether electrical stimulation of the eighth cranial nerve also affects vestibular functions and determine if the stimulaton changes postural stability and created compensations.

DETAILED DESCRIPTION:
The patient undergoes a comprehensive examination of posture, stability of standing in 10 different conditions, stability of standing with sound stimulation, visual vertical examination and evaluation of the current mental state and subjective perception of difficulties through a questionnaire survey. All will be repeated four times at regular intervals. The investigators examine the patient before the surgery, 1 day after the surgery, 2-3 weeks afer it when the surgeons expect a stabilization of the postoperative condition, and with a gap of at least 6 months after the surgery, when the patient has already completed the adjustment of the speech processor and the compensation has been already created. Standing stability will be evaluated for 30 s in 10 different conditions with eyes open/closed eyes, with or without the foam, in a neutral head position/with an extended head, in a supine standing position/in tandem. The examination room include audio technology for playing sound, thanks to which the examinators can also assess the influence of sound perception and cognitive processes on maintaining stability during the measurement. The investigators will perform the stimulation while standing without visual control on the foam in 6 different sound conditions. With the speech processor on and off, with the white noise, spoken words in Czech language, for the patient completly foreign language (Finnish, or Chinese) and focused listening (simulated dual tasking) with control question at the end of the stimulation. Another method will be the examination of the perception of the subjective visual vertical. This is considered as a sensitive tool to detect asymmetric function of the labyrinths. The testing is in sitting position and controlled by a joystick move a straight line projected on a widescreen 2 meters infront of the participant. The examination is in static and dynamic mode, when during the dynamic examination, optokinetic stimulation occurs, which makes difficult to determine the vertical position. Standardized questionnaires will be used to evaluate subjectively perceived difficulties, quality of life and occurrence of psychological problems related to postural instability and underwent surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients who meet the demanding indication criteria for cochlear implantation (include an ENT examination, audiometry, neurological examination, examination by a clinical speech therapist and by a psychologist and CT examination of the temporal bones) also meet the conditions for inclusion into the study

Exclusion Criteria:

* the presence of diseases of the load-bearing joints of the limbs
* the presence of diseases of peripheral nervous system or muscle disease
* the presence of disease of vision which would make visual fixation impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: working age candidates who are coming for cochlear implantation from all of the country
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-01-11 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
In patients with the cochlear implant there are changes in the function of the vestibular system, specifically in sway path. | Pre operative - baseline, than 1st day after surgery, 2-3 weeks after surgery and than at least 6 months after the surgery
  Compare of the result parameters from posturography as the sway path in mm in total, AP and ML directions. Testing before (baseline) and after the surgery in the same patient.
In patients with the cochlear implant there are changes in the function of the vestibular system, specifically in sway area. | Pre operative - baseline, than 1st day after surgery, 2-3 weeks after surgery and than at least 6 months after the surgery
  Compare of the result parameters from posturography as the sway area in mm*2 in total, AP and ML directions. Testing it before (baseline) and after the surgery in the same patient.
In patients with the cochlear implant there are changes in the function of the vestibular system, specifically in the sway velocity. | Pre operative - baseline, than 1st day after surgery, 2-3 weeks after surgery and than at least 6 months after the surgery
  Compare of the result parameters from posturography as the sway velocity in m/s in total, AP and ML directions. Testing before (baseline) and after the surgery in the same patient.

SECONDARY OUTCOMES:
In patients with the cochlear implant there are changes in the function of the vestibular system, specifically in the subjective visual vertical. | Pre operative - baseline, than 1st day after surgery, 2-3 weeks after surgery and than at least 6 months after the surgery
  Evaluate the measurement of subjective visual vertical in angular degrees. If it follows the normal values or if the deviation from vertical is higher than 2°. Testing before (baseline) and after the surgery in the same patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rehabilitation and Sports Medicine, 2nd Medical Faculty, Charles University and University Hospital Motol, Prague, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Koutna S, Kalitova P, Jerabek J, Slaby K, Kucerova K, Boucek J, Cakrt O. Comparison of postural control and space perception outcomes between robotic and conventional cochlear implantation in adults. Eur Arch Otorhinolaryngol. 2024 Jul;281(7):3839-3843. doi: 10.1007/s00405-024-08664-3. Epub 2024 Jun 2. PMID 38825603